CLINICAL TRIAL: NCT04705831
Title: A Randomized, Double Blind, Placebo Controlled, Cross-Over, Proof-of-Concept Study to Evaluate the Benefit of RUCONEST (C1 Esterase Inhibitor [Recombinant]) in Improving Neurological Symptoms in Post-SARS-CoV-2 Infection
Brief Title: Study to Evaluate the Benefit of RUCONEST in Improving Neurological Symptoms in Post COVID-19 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IMMUNOe Research Centers (Industry)
Responsible Party: Principal Investigator, Isaac Melamed, MD, Principal Investigator, IMMUNOe Research Centers
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IIS202001-Neuroimmune
Record Dates: First submitted 2021-01-07; First posted 2021-01-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2021-01

CONDITIONS: Post-Viral Fatigue Syndrome; Post-Viral Disorder (Disorder); Covid19
Keywords: Post-COVID Symptoms; Post-Viral Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic; COVID-19 | interventions — conestat alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- RUCONEST (Active Comparator): IV Ruconest
  Interventions: Drug: Ruconest
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Ruconest

INTERVENTIONS:
Drug: Ruconest — C1 Esterase Inhibitor

SUMMARY:
Randomized, Double Blind, Placebo Controlled, Proof-of-Concept Study to Evaluate the Benefit of RUCONEST in Improving Neurological Symptoms in Post-SARS-CoV-2 Infection.

DETAILED DESCRIPTION:
This study will last approximately 19 weeks including 16 infusions total, each one week apart. This is to help patients that have developed "Post-Viral Fatigue Syndrome" which can include symptoms such as: extreme fatigue, lost of taste, brain fog, and/or seizures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older, male or female
2. Previous confirmed diagnosis of SARS-CoV-2
3. Experiencing SARS-CoV-2 post-viral fatigue syndrome 4 weeks after recovery for SARS-CoV-2
4. Experiencing neurological symptoms including fatigue
5. Willing to comply with all aspects of the protocol, including blood draws
6. Patient is able to understand and fully participate in the activities of the study and the consent in accordance with guidelines
7. Female patients of childbearing potential who are sexually active must be willing to use an acceptable form of contraception. Acceptable forms of contraception are defined as those with a failure rate of < 1% when properly applied and include: a combination pill, some intra-uterine devices, and a sterilized partner in a stable relationship. Female patients must not be pregnant, planning to become pregnant, or be actively breastfeeding through the entire period.

Exclusion Criteria:

1. Receiving any form of C1-INH therapy either acute or prophylactic treatment
2. History or suspicion of allergy to rabbits
3. Neurological conditions related to injury
4. Neuropathy related to diabetes
5. Participants who are pregnant or lactating
6. Largely incapacitated or bed ridden
7. Currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study or have discontinued with 30 days of study entry from any other clinical study involving an investigational product
8. Patients who, in the investigator's opinion, might not be suitable for the trial for safety reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Neuropsychological Measures (BRIEF-A) | Week 0
  Behavior Rating Inventory of Executive Function- Adult (BRIEF-A)
Neuropsychological Measures (BRIEF-A) | Week 9
  Behavior Rating Inventory of Executive Function- Adult (BRIEF-A)
Neuropsychological Measures (BRIEF-A) | Week 17
  Behavior Rating Inventory of Executive Function- Adult (BRIEF-A)
Neuropsychological Measures (RBANS) | Week 0
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Neuropsychological Measures (RBANS) | Week 9
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Neuropsychological Measures (RBANS) | Week 17
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Neuropsychological Measures (BDI II) | Week 0
  Beck Depression Inventory II (BDI II)
Neuropsychological Measures (BDI II) | Week 9
  Beck Depression Inventory II (BDI II)
Neuropsychological Measures (BDI II) | Week 17
  Beck Depression Inventory II (BDI II)
Neuropsychological Measures (MoCA) | Week 0
  Montreal Cognitive Assessment (MoCA)
Neuropsychological Measures (MoCA) | Week 9
  Montreal Cognitive Assessment (MoCA)
Neuropsychological Measures (MoCA) | Week 17
  Montreal Cognitive Assessment (MoCA)
Patient-Rate Questionnaires (FSS) | Week 0
  Fatigue Severity Scale (FSS)
Patient-Rate Questionnaires (FSS) | Week 5
  Fatigue Severity Scale (FSS)
Patient-Rate Questionnaires (FSS) | Week 9
  Fatigue Severity Scale (FSS)
Patient-Rate Questionnaires (FSS) | Week 14
  Fatigue Severity Scale (FSS)
Patient-Rate Questionnaires (FSS) | Week 17
  Fatigue Severity Scale (FSS)
Patient-Rate Questionnaires (MIDAS) | Week 0
  Migraine Disability Assessment (MIDAS)
Patient-Rate Questionnaires (MIDAS) | Week 5
  Migraine Disability Assessment (MIDAS)
Patient-Rate Questionnaires (MIDAS) | Week 9
  Migraine Disability Assessment (MIDAS)
Patient-Rate Questionnaires (MIDAS) | Week 14
  Migraine Disability Assessment (MIDAS)
Patient-Rate Questionnaires (MIDAS) | Week 17
  Migraine Disability Assessment (MIDAS)
Patient-Rate Questionnaires (HIT) | Week 0
  Headache Impact Scale (HIT)
Patient-Rate Questionnaires (HIT) | Week 5
  Headache Impact Scale (HIT)
Patient-Rate Questionnaires (HIT) | Week 9
  Headache Impact Scale (HIT)
Patient-Rate Questionnaires (HIT) | Week 14
  Headache Impact Scale (HIT)
Patient-Rate Questionnaires (HIT) | Week 17
  Headache Impact Scale (HIT)
Patient-Rate Questionnaires (Activities) | Week 0
  Activities of Daily Living Sliding Scale and Questionnaire
Patient-Rate Questionnaires (Activities) | Week 5
  Activities of Daily Living Sliding Scale and Questionnaire
Patient-Rate Questionnaires (Activities) | Week 9
  Activities of Daily Living Sliding Scale and Questionnaire
Patient-Rate Questionnaires (Activities) | Week 14
  Activities of Daily Living Sliding Scale and Questionnaire
Patient-Rate Questionnaires (Activities) | Week 17
  Activities of Daily Living Sliding Scale and Questionnaire
Patient-Rate Questionnaires (SF) | Week 0
  SF McGill Pain Questionnaire
Patient-Rate Questionnaires (SF) | Week 5
  SF McGill Pain Questionnaire
Patient-Rate Questionnaires (SF) | Week 9
  SF McGill Pain Questionnaire
Patient-Rate Questionnaires (SF) | Week 14
  SF McGill Pain Questionnaire
Patient-Rate Questionnaires (SF) | Week 17
  SF McGill Pain Questionnaire
Patient-Rate Questionnaires (GSRS) | Week 0
  Gastrointestinal Symptoms Rating Scale (GSRS)
Patient-Rate Questionnaires (GSRS) | Week 5
  Gastrointestinal Symptoms Rating Scale (GSRS)
Patient-Rate Questionnaires (GSRS) | Week 9
  Gastrointestinal Symptoms Rating Scale (GSRS)
Patient-Rate Questionnaires (GSRS) | Week 14
  Gastrointestinal Symptoms Rating Scale (GSRS)
Patient-Rate Questionnaires (GSRS) | Week 17
  Gastrointestinal Symptoms Rating Scale (GSRS)
Patient-Rate Questionnaires (SF-36) | Week 0
  SF-36
Patient-Rate Questionnaires (SF-36) | Week 5
  SF-36
Patient-Rate Questionnaires (SF-36) | Week 9
  SF-36
Patient-Rate Questionnaires (SF-36) | Week 14
  SF-36
Patient-Rate Questionnaires (SF-36) | Week 17
  SF-36
Neurological Exam (0) | Week 0
  Complete neurological examination
Neurological Exam (9) | Week 9
  Complete neurological examination
Neurological Exam (17) | Week 17
  Complete neurological examination
Immunological Biomarkers (Toll) | Week 1
  Toll Like Receptor Function Assay
Immunological Biomarkers (Toll) | Week 9
  Toll Like Receptor Function Assay
Immunological Biomarkers (Toll) | Week 17
  Toll Like Receptor Function Assay
Immunological Biomarkers (GAD) | Week 1
  GAD-65
Immunological Biomarkers (GAD) | Week 9
  GAD-65
Immunological Biomarkers (GAD) | Week 17
  GAD-65
Immunological Biomarkers (Com) | Week 1
  Complement Panel (C4, C1-INH, C1-INH Function)
Immunological Biomarkers (Com) | Week 9
  Complement Panel (C4, C1-INH, C1-INH Function)
Immunological Biomarkers (Com) | Week 17
  Complement Panel (C4, C1-INH, C1-INH Function)
Immunological Biomarkers (Ig) | Week 1
  Immunoglobulins-Quantitative (IgA, IgE, IgG, IgM)
Immunological Biomarkers (Ig) | Week 9
  Immunoglobulins-Quantitative (IgA, IgE, IgG, IgM)
Immunological Biomarkers (Ig) | Week 17
  Immunoglobulins-Quantitative (IgA, IgE, IgG, IgM)
Immunological Biomarkers (IgG) | Week 1
  Immunoglobulins G, Subclasses (1-4)
Immunological Biomarkers (IgG) | Week 9
  Immunoglobulins G, Subclasses (1-4)
Immunological Biomarkers (IgG) | Week 17
  Immunoglobulins G, Subclasses (1-4)
Immunological Biomarkers (TH/TH) | Week 1
  TH1/TH2 Cytokine Levels
Immunological Biomarkers (TH/TH) | Week 9
  TH1/TH2 Cytokine Levels
Immunological Biomarkers (TH/TH) | Week 17
  TH1/TH2 Cytokine Levels

CONTACTS AND LOCATIONS:
Locations (1):
- IMMUNOe Research Centers, Centennial, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Melamed I, Buckley C, Bayko ME, Williams JL, Or-Geva N. Does C1 esterase inhibitor play a role in post COVID-19 neurological symptoms? A randomized, double-blind, placebo-controlled, crossover, proof-of-concept study. Front Neurol. 2025 Nov 6;16:1523814. doi: 10.3389/fneur.2025.1523814. eCollection 2025. PMID 41281561